CLINICAL TRIAL: NCT05545046
Title: A Predictive Model for Pain After Transarterial Chemoembolization
Brief Title: Predictive Model for Pain After TACE
Status: Completed | Type: Observational
Sponsor: Yantai Yuhuangding Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-406
Record Dates: First submitted 2022-09-14; First posted 2022-09-19 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 16 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main aim of this study was to analyze the risk factors that helped to predict the pain after transarterial chemoembolization (TACE).This was a prospective observational study enrolled all hepatocellular carcinoma (HCC) patients undergoing TACE in our hospital. Pain score at rest was assessed after TACE by the patients themselves using a Visual Analogue Scale (VAS). Independent variables such as age, gender, tumor location, tumor size and number, drug delivery method and presence of portal vein tumor thrombosis (PVTT) were recorded and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of HCC was confirmed either histologically or based on consistent findings obtained from at least two imaging techniques.

Exclusion Criteria:

* patients aged < 18 year
* significant heart or lung dysfunction
* use of additional analgesics to relieve pain during TACE
* cognitive impairment
* use of psychiatric medications
* drug or alcohol abuse

Ages: 34 Years to 87 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A diagnosis of HCC was confirmed either histologically or based on consistent findings obtained from at least two imaging techniques.
Sampling Method: Non-Probability Sample
Enrollment: 228 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | 0 hour after TACE by the patients themselves using a Visual Analogue Scale (VAS)
  After local anesthesia with an injection of 10 mL of 2% lidocaine, all the patients enrolled in this study received percutaneous femoral artery puncture. An arterial catheter was inserted into the femoral artery and subsequently placed in the hepatic artery. Then, a conventional TACE or a DEB-TACE procedure was performed. After TACE, all patients received supportive treatment including antiemetics, liver protection, non-steroidal anti-inflammatory drugs.
Visual Analogue Scale (VAS) | 2 hour after TACE by the patients themselves using a Visual Analogue Scale (VAS)
  After local anesthesia with an injection of 10 mL of 2% lidocaine, all the patients enrolled in this study received percutaneous femoral artery puncture. An arterial catheter was inserted into the femoral artery and subsequently placed in the hepatic artery. Then, a conventional TACE or a DEB-TACE procedure was performed. After TACE, all patients received supportive treatment including antiemetics, liver protection, non-steroidal anti-inflammatory drugs.
Visual Analogue Scale (VAS) | 4 hour after TACE by the patients themselves using a Visual Analogue Scale (VAS)
  After local anesthesia with an injection of 10 mL of 2% lidocaine, all the patients enrolled in this study received percutaneous femoral artery puncture. An arterial catheter was inserted into the femoral artery and subsequently placed in the hepatic artery. Then, a conventional TACE or a DEB-TACE procedure was performed. After TACE, all patients received supportive treatment including antiemetics, liver protection, non-steroidal anti-inflammatory drugs.
Visual Analogue Scale (VAS) | 6 hour after TACE by the patients themselves using a Visual Analogue Scale (VAS)
  After local anesthesia with an injection of 10 mL of 2% lidocaine, all the patients enrolled in this study received percutaneous femoral artery puncture. An arterial catheter was inserted into the femoral artery and subsequently placed in the hepatic artery. Then, a conventional TACE or a DEB-TACE procedure was performed. After TACE, all patients received supportive treatment including antiemetics, liver protection, non-steroidal anti-inflammatory drugs.
Visual Analogue Scale (VAS) | 12 hour after TACE by the patients themselves using a Visual Analogue Scale (VAS)
  After local anesthesia with an injection of 10 mL of 2% lidocaine, all the patients enrolled in this study received percutaneous femoral artery puncture. An arterial catheter was inserted into the femoral artery and subsequently placed in the hepatic artery. Then, a conventional TACE or a DEB-TACE procedure was performed. After TACE, all patients received supportive treatment including antiemetics, liver protection, non-steroidal anti-inflammatory drugs.
Visual Analogue Scale (VAS) | 24 hour after TACE by the patients themselves using a Visual Analogue Scale (VAS)
  After local anesthesia with an injection of 10 mL of 2% lidocaine, all the patients enrolled in this study received percutaneous femoral artery puncture. An arterial catheter was inserted into the femoral artery and subsequently placed in the hepatic artery. Then, a conventional TACE or a DEB-TACE procedure was performed. After TACE, all patients received supportive treatment including antiemetics, liver protection, non-steroidal anti-inflammatory drugs.

CONTACTS AND LOCATIONS:
Locations (1):
- Yuhuangding Hospital, Yantai, Shandong, China